CLINICAL TRIAL: NCT04950049
Title: The Effect of Dilution With Glucose and Prolonged Injection Time on Dexamethasone-induced Perineal Irritation
Brief Title: The Effect of Dilution and Prolonged Injection Time on Dexamethasone-induced Perineal Irritation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Zhangyonghai02
Record Dates: First submitted 2020-10-23; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Adverse Effect
Keywords: Dexamethasone 21-phosphate; Pain; Pruritus; Glucose
MeSH Terms: conditions — Pain; Pruritus | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2 ml dexamethasone (5 mg/ml) (Active Comparator): 50 patients receive 2 ml dexamethasone (5 mg/ml) , the injection time of dexamethasone was less than 2s.
  Interventions: Drug: Dexamethasone
- 5 ml dexamethasone (2mg/ml) (Experimental): 50 patients receive 5 ml dexamethasone (2mg/ml) diluted with 5% glucose, the injection time of dexamethasone was 30s.
  Interventions: Other: Diluted dexamethasone 5ml
- 10 ml dexamethasone (1mg/ml) (Experimental): 50 patients receive 10 ml dexamethasone (1mg/ml) diluted with 5% glucose, the injection time of dexamethasone was 30s.
  Interventions: Other: Diluted dexamethasone 10ml
- 20 ml dexamethasone (0.5mg/ml) (Experimental): 50 patients receive 20 ml dexamethasone (0.5mg/ml) diluted with 5% glucose, the injection time of dexamethasone was 30s.
  Interventions: Other: Diluted dexamethasone 20ml

INTERVENTIONS:
Drug: Dexamethasone — receive 2ml dexamethasone (5mg/ml)
  Arms: 2 ml dexamethasone (5 mg/ml)
Other: Diluted dexamethasone 5ml — receive 5ml dexamethasone (2mg/ml) diluted with 5% glucose
  Arms: 5 ml dexamethasone (2mg/ml)
Other: Diluted dexamethasone 10ml — receive 10ml dexamethasone (1mg/ml) diluted with 5% glucose
  Arms: 10 ml dexamethasone (1mg/ml)
Other: Diluted dexamethasone 20ml — receive 20ml dexamethasone (0.5mg/ml) diluted with 5% glucose
  Arms: 20 ml dexamethasone (0.5mg/ml)

SUMMARY:
The purpose of this study is to investigate the efficacy of dilution with glucose and prolonged injection time on dexamethasone 21-phosphate induced perineal irritation (include pian and pruritus).

DETAILED DESCRIPTION:
Dexamethasone is a synthetic glucocorticoid, which may cause perineal irritation when given intravenously. The major clinical manifestations are pruritus and pain，and the incidence vary between 38%-71%. Some patients undergo spontaneous remission, while others develop into severe pain or pruritus. In clinical practice, dexamethasone is always diluted with glucose in many cases, but diluted dexamethasone in relieving dexamethasone induced perineal irritation has not been studied yet. The aim of this study was to investigate the efficacy of dilution with glucose on dexamethasone induced perineal irritation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* ASA physical status I-II

Exclusion Criteria:

* On regular use of analgesic
* Contraindication or allergy to steroid or glucose
* Drug or alcohol abuse
* Diagnosed with paresthesia or mental diseases
* Communication disorders
* Pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dexamethasone-induced perineal irritation | During the first 3 min period after the injection of dexamethasone
  The investigators record the number of cases of dexamethasone-induced perineal irritation (pain or pruritus) and calculate the incidence

SECONDARY OUTCOMES:
Duration of perineal irritation | After the injection of dexamethasone, up to 5 minutes
  If perineal irritation occurs, the investigators will record its duration
The severity of perineal irritation | After the injection of dexamethasone, up to 5 minutes
  If perineal irritation occurs, the investigators will assess its severity by using Visual Analogue Scale (the minimum is 0 and the maximum is 10, and the higher scores mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Yonghai Zhang, Principal Investigator — General Hospital of Ningxia Medical University

IPD SHARING:
Plan to Share IPD: Undecided